CLINICAL TRIAL: NCT01865292
Title: A Randomised, Double-Blind, Single Dose, Six-Period Cross-over Dose Response Trial Comparing the Pharmacodynamics and Pharmacokinetics of Insulin 454 With Insulin Glargine in Subjects With Type 1 and Type 2 Diabetes
Brief Title: Comparing the Pharmacodynamics and Pharmacokinetics of Explorative Formulation of Insulin Degludec With Insulin Glargine in Subjects With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1719; 2006-001915-31 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec (Experimental)
  Interventions: Drug: insulin degludec
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Three single doses administrated subcutaneously (s.c., under the skin) on three separate dosing visits. Dose will vary when administered to subjects with type 1 and type 2 diabetes, respectively.
  Arms: Insulin degludec
Drug: insulin glargine — Three single doses administrated subcutaneously (s.c., under the skin) on three separate dosing visits. Dose will vary when administered to subjects with type 1 and type 2 diabetes, respectively.
  Arms: Insulin glargine

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the pharmacodynamics (the effect of the investigated drug on the body) and pharmacokinetics (the exposure of the trial drug in the body) of insulin degludec (insulin 454), an explorative formulation, not similar to the proposed commercial formulation, with insulin glargine in subjects with type 1 and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Glycosylated haemoglobin (HbA1c) below or equal to 10 procent based on central laboratory results
* Specific inclusion criteria for subject with type 1 diabetes:
* Diagnosed with type 1 diabetes mellitus and treated with insulin for at least 12 months prior to screening
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)
* Specific inclusion criteria for subject with type 2 diabetes:
* Diagnosed with type 2 diabetes mellitus for at least 12 months prior to screening
* Treated with insulin for the past 3 months prior to screening
* Body Mass Index (BMI) between 22.0 and 35.0 kg/ m^2 (both inclusive)

Exclusion Criteria:

* Subject with a history of significant multiple drug allergies or with a known allergy or suspected allergy to the trial product or any medicine chemically related to the trial product,as judged by the Investigator.
* Subject with a history of or presence of cancer
* Any condition that the Investigator and/or Sponsor feels would interfere with study
* Specific exclusion criteria for subject with type 2 diabetes:
* Therapy with oral antidiabetic drugs within the past 3 months prior to screening

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | 0-24 hours after dosing

SECONDARY OUTCOMES:
Area under the insulin degludec/insulin glargine curve | 0-96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com